CLINICAL TRIAL: NCT03284736
Title: Effects of Guided Tissue Regeneration on the Healing of Through & Through Periradicular Lesions: A Randomized Controlled Study
Brief Title: Guided Tissue Regeneration in the Healing of Through and Through Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pragnesh endo
Record Dates: First submitted 2017-09-08; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Periapical Lesions

STUDY DESIGN:
Intervention Model Description: A total number of 15 patients in each group were selected. Patients were randomly allocated by computer program into two group. Clinical and radiographic examinations were performed every 3, 6 and 12 months by assessing the same parameters as baseline except that PD, CAL, and GMP were measured until 12 months. Routine examination procedure were used to evaluate any evidence of signs and/or symptoms. Jig radiographs were taken at 3, 6 and 12th month of follow up. Inter and intra observation of data will be analyzed by distribution of data. Categorical data will be analyzed by chi square test. Regression analysis will be done to observe any association between independent and dependent variables. Interobserver/intraobserver reliability with cohen kappa analysis.
Who Masked: Participant, Investigator
Masking Description: Both the participant and primary investigator are blinded in the study until whole surgical procedure is completed and before suturing the flap.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periapical surgery with membrane (Experimental): After retrofilling of teeth with MTA , defect was covered with collagen resorbable membrane.
  healiguide collagen type 1 resorbable membrane covering the defect by extending 2-3 mm in every direction.
  Interventions: Procedure: Resorbable membrane
- Periapical surgery without membrane. (Active Comparator): After retrofilling of teeth with MTA, flap was closed without application of collagen resorbable membrane.
  Interventions: Procedure: periapical surgery without membrane

INTERVENTIONS:
Procedure: Resorbable membrane
  Other Names: Healiguide collagen type 1 resorbable membrane
  Arms: Periapical surgery with membrane
Procedure: periapical surgery without membrane — after removing pathology and retro-filling the tooth /teeth wit MTA the defect area is left as it is and flap is closed without resorbable membrane.
  Arms: Periapical surgery without membrane.

SUMMARY:
Study Title: Effects of Guided Tissue Regeneration on the Healing of Through & Through Periradicular Lesions - A Randomized Controlled Study

Rationale: Through and through defects found to be difficult to heal without GTR intervention. Various studies has been done either with graft or without graft but no randomized controlled trial has been done on resorbable membrane(GTR) in through and through lesion.

Aim & Objectives: To evaluate the effect of resorbable collagen membrane in the healing of through & through lesion.

Setting: Study was conducted in Post Graduate Institute Of Dental Sciences, Rohtak in the department of Conservative Dentistry & Endodontics.

Study Design: Randomized Controlled Trial

Time Frame: March 2016 to October 2017

Population / Participants: Patients of age 16 years (male/female) and above were enrolled in the study.

Inclusion Criteria: Patients of age 16 years and above, -ve response to vitality test, failed previous root canal treatment with purulent discharge, failed previous surgery, recurrent episode of purulent discharge.

Exclusion Criteria: Unrestorable tooth, fractured /perforated roots, serious medical illness, smokers, pregnant females and lactating mothers, grade 3 mobile teeth, the need for antibiotic prophylaxis prior to dental care.

Sample size: 30 patients (15 patients in each group)

Methods: Clinically and radiographically diagnosis of lesion, vitality check by EPT, preoperative evaluation by bleeding on probing, clinical attachment level, gingival marginal position & pocket depth. Surgical procedures will be carried out under operating microscope with 8 × 16 magnification by following standardized treatment methods.

Outcome measures: Follow up of patients were carried out at 3, 6, 9 & 12 months and outcome measures were compared with same method done pre operatively and described as Complete healing, incomplete healing (scar tissue), uncertain healing, unsatisfactory healing (failure).

Statistical method: Data will be analyzed with suitable statistics method.

DETAILED DESCRIPTION:
The research process was carried out in the Department Of Conservative Dentistry and Endodontics, Post Graduate Institute of Dental Sciences, Rohtak. Patients with through and through periradicular lesions diagnosed radiographically and clinically were be included in the study.

INCLUSION CRIETERIA :-

1. Patients of age 16 years and above with a clinical & radiographic diagnosis of through and through periradicular lesion.
2. Negative response to vitality test with radiographic evidence of periapical rediolucencies.
3. Failed previous root canal treatment with purulent discharge and radiographic evidence of periapical pathology.
4. Failed previous surgery with persistent bony lesion.
5. Recurrent episode of purulent discharge and adequate final restoration with no clinical evidence of coronal leakage.

EXCLUSION CRIETERIA :-

1. Unrestorable tooth
2. Fractured /perforated roots
3. Serious medical illness (uncontrolled/poorly controlled diabetes, unstable or life threatening conditions or requiring antibiotic prophylaxis)
4. Smokers
5. Pregnant females and lactating mothers
6. Grade 3 mobile teeth
7. The need for antibiotic prophylaxis prior to dental care

Baseline parameters --

Endodontic evaluation - Pulp sensibility testing was performed with a combination of heat test (heated gutta-percha), cold test (Endo-Frost, Coltene Whale dent) and electric pulp test (Digitestz D626D, Parkell electronics, New York). Teeth not responding to both thermal and electric test were considered non vital.

Radiographic evaluation - Radiographs with paralleling cone technique was taken at baseline and at subsequent appointments at standardized exposure parameters (70kvp, 3.5mAs, and 0.2 seconds).

Clinical Periodontal Evaluation - The following clinical parameters were evaluated at baseline and at subsequent follow up appointments in the test tooth and the contra lateral normal tooth in the same patient.

1. Bleeding on probing - The presence or absence of bleeding following pocket probing were recorded at 6 sites per tooth - mesiobuccal, buccal, distobuccal, mesiolingual, midlingual, distolingual. This assessment was done in full mouth.
2. Probing pocket depth (PPD) - Probing depth was measured as the distance from the gingival margin to the base of the clinical pocket. The probing depth measurements was assessed using a calibrated manual periodontal Williams 0 probe. The probe was inserted with a firm, gentle pressure to the bottom of the pocket and maintained parallel to the vertical axis of the tooth. Measurements were noted at 6 sites per tooth- mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual. Measurements will be rounded to the nearest whole millimeter.
3. Clinical Attachment Level (CAL) - Clinical Attachment Level was measured as the distance between the base of the clinical pocket and a fixed point on the crown, the cementoenamel junction (CEJ). Measurements were made at 6 sites per tooth- mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual using wiliiams 0 probe. Measurements were rounded to the nearest whole millimeter. The mean CAL over all examined surfaces were calculated.
4. Gingival marginal level/position from CEJ was measured.Radiographic examination was performed at 0, 3, 6, 9 and 12 months by using Rinn ( XCP instruments, Elgin, IL ) paralleling technique digitized by using Kodak RVG 6000 ( Kodak Digital Radiographic System, Pt Husada Intra Care, Banten, Indonesia ).

SAMPLE SIZE

A total number of 15 patients in each group were selected. Sample size was determined by calculating the difference of success rate between the previous studies of GTR procedures.

1. Test Group: 15 Non vital teeth having through and through periradicular lesion diagnosed clinically and radiographically first treated with conventional endodontic treatment. After follow up of one month if no improvement found clinically and radiographically then apical surgery was carried out using guided tissue regeneration in patients.
2. Control Group: 15 Non vital teeth having through and through periradicular lesion diagnosed clinically and radiographically first treated with conventional endodontic treatment. After follow up of one month if no improvement found clinically and radiographically then apical Surgery was carried out without using guided tissue regeneration.

RANDOMIZATION

Patients were randomly allocated by computer program [ Random Allocation Software (http://www.msaghaei.com/Softwares/dnld/RA.zip) ] into two group. Group I=Collagen membrane group (MG), group II=Control group (CG).

SURGICAL TECHNIQUE:

With the exception of incisions, flap elevation and suturing, all surgical procedures was performed under operating microscope in an operating room under 8x to 16x magnification.

The full thickness (mucoperiosteal flap) was reflected under aseptic condition by the following technique

1. Preoperative mouth rinse with 0.2% chlorhexidine mouthwash was used.
2. Local anaesthesia with lidocaine 2% with epinephrine 1:80,000 was achieved.
3. Buccal intrasulcular incision was given up to the alveolar crest including one tooth mesial to the lesion & two teeth distal to the lesion, using no.15 blade on handle.
4. Mesial and distal vertical releasing incision were given.
5. Full thickness flap was gently reflected towards the apical area by periosteal elevator. The flap was frequently irrigated with sterile saline to prevent dehydration of periosteal surface.
6. After complete elevation of the flap, debridement (periradicular curettage -enucleation) of the bony lesion was performed. For additional hemostasis during surgery, cotton pellets soaked in 0.1% epinephrine was applied topically as required.
7. A 2-3mm root tip with a 0º to 10º bevel angle was sectioned with cylindrical surgical carbide burs at high speed with sterile water coolant.
8. Root end preparations extending 3mm into the canal space along the long axis of the root was made by using a piezoelectric ultrasonic system with double angled Retrotips coated with Diamond abrasives.
9. Isthmuses, fins, and other significant anatomic irregularities were identified in high magnification and was treated with the ultrasonic instruments. Then the resected root surfaces was stained with methylene blue and were inspected with micromirrors under high magnification of 24x to examine the cleanliness of the root end preparation and detect any other overlooked anatomic details.
10. Root end filling were with mineral trioxide aggregrate (MTA). The adaptation of the filling material to the canal apical walls was confirmed with the aid of an operating microscope at high magnification.
11. After MTA retrofilling in the test group Collagen membrane was applied on buccal side and in the control group nothing was apllied and flap will be closed with 4-0 reverse cutting black silk suture.

RESORBABLE COLLAGEN MEMBRANE:

Bioabsorbable membranes are composed of a wide variety of materials including collagen, polylactic acid, polyurethane, polyglactin 910, acellular dermal matrix, dura mater, chitosan, periosteum, and calcium sulfate. The most common material is collagen, which can be modified through various collagen cross-linking processing techniques to vary the resorption rate.

Numerous studies have shown bioabsorbable membranes to be effective at promoting regeneration in both endodontic and periodontal defects. Because alveolar bone and the periodontal ligament contain collagen, using a collagen membrane might impart some additional advantages for GTR purposes by augmenting its native properties.

Collagen facilitates hemostasis and therefore wound stability by promoting platelet aggregation in addition to promoting fibroblast migration, which could accelerate wound closure. After inspecting the root end filled teeth with microscope and radiographically the defect will be covered with resorbable collage membrane.

Postoperative instructions:

Care must be taken not to over compress the area. patient should rinse with an appropriate antimicrobial agent of the clinician's choice (chlorhexidine glucoanate) twice daily for two weeks. patient should avoid brushing the area for 2 weeks from the surgery date, avoid flossing for 4 weeks from surgery date. following the first 2 weeks from surgery for the next 3 weeks it is recommended to brush the area only with soft brush.

Post - Operative Follow-Up:

Clinical and radiographic examinations were performed every 3, 6 and 12 months by assessing the same parameters as baseline except that PD, CAL, and GMP were not measured until 12 months. Routine examination procedure was used to evaluate any evidence of signs and/or symptoms.

Radiographic evaluations:

Jig radiographs will be taken at 3, 6 and 12th month of follow up. Radiographic healing will be assessed by the criteria as below.

1. Complete healing, defined by re-establishment of the lamina dura
2. Incomplete healing (scar tissue)
3. Uncertain healing
4. Unsatisfactory healing (failure)

Processing Of Data:

Inter and intra observation of data will be analyzed by distribution of data. Categorical data will be analyzed by chi square test. Regression analysis will be done to observe any association between independent and dependent variables. Interobserver/intraobserver reliability with cohen kappa analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age 16 years and above with a clinical & radiographic diagnosis of through and through periradicular lesion.
2. Negative response to vitality test with radiographic evidence of periapical rediolucencies.
3. Failed previous root canal treatment with purulent discharge and radiographic evidence of periapical pathology.
4. Failed previous surgery with persistent bony lesion.
5. Recurrent episode of purulent discharge and adequate final restoration with no clinical evidence of coronal leakage.

Exclusion Criteria:

1. Unrestorable tooth
2. Fractured /perforated roots
3. Serious medical illness (uncontrolled/poorly controlled diabetes, unstable or life threatening conditions or requiring antibiotic prophylaxis)
4. Smokers
5. Pregnant females and lactating mothers
6. Grade 3 mobile teeth
7. The need for antibiotic prophylaxis prior to dental care

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Change in periapical radiolucency by radiograph 1. Complete healing, 2. Incomplete healing 3. Uncertain healing 4. Unsatisfactory healing | Baseline to 1 year
  Healing of the lesion will be checked at 3 months interval up to 1 year with the help of software CDR DICOM. At the end of 1 year this reduction in the pathology of lesion will be categorized as complete, incomplete, uncertain, unsatisfactory.
  Clinical and radiographic examinations will be performed every 3, 6 and 12 months by assessing the same parameters as baseline except that PD, CAL, and GMP will not measured until 12 months.
  Radiographic evaluations Jig radiographs will be taken at 3, 6 and 12th month of follow up.

SECONDARY OUTCOMES:
Clinical attachment level | Baseline to 1 year
  At the end of 1 year clinical attachment level will be checked of involved teeth.
Probing depth | Baseline to 1 year
  At the end of 1 year probing depth and will be checked of involved teeth.

IPD SHARING:
Plan to Share IPD: Yes